CLINICAL TRIAL: NCT05415774
Title: Combined Deep Brain Stimulation of the Substantia Nigra Pars Reticulata and of the Subthalamic Nucleus for Unresponsive Freezing of Gait in Parkinson's Disease: a Pilot Cross-over Study
Brief Title: Combined Deep Brain Stimulation in Parkinson's Disease
Acronym: SCP-FOG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: RC31/21/0609
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2023-12

CONDITIONS: Parkinson Disease
Keywords: freezing of gait; deep brain stimulation; combined deep brain stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Single center, randomized, three one-month periods, six sequences, cross-over, double blind, study to evaluate the effect of 2 innovative settings of DBS combining the stimulation of STN and SNr, vs. a standard (S) stimulation, on FoG, in PD patients with DBS with severe FoG.
  the sequence of different stimulation parameters will be randomized and not the treatment Each patient receives the three treatments (S, C1 and C2)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- S Stimulation (Active Comparator): Standard STN DBS defined as high frequency at 130Hz stimulation
  Interventions: Device: 1 : S-C1-C2; Device: 2 : S-C2-C1; Device: 3 : C1 - S - C2; Device: 4 : C1 -C2 - S; Device: 5 : C2 - S - C1; Device: 6 : C2 - C1 - S
- C1 Stimulation (Experimental): Combined high frequency stimulation of the STN and SNr using an interleaved pulses at 125Hz
  Interventions: Device: 1 : S-C1-C2; Device: 2 : S-C2-C1; Device: 3 : C1 - S - C2; Device: 4 : C1 -C2 - S; Device: 5 : C2 - S - C1; Device: 6 : C2 - C1 - S
- C2 Stimulation (Experimental): Combined low frequency stimulation of the SNr at 60Hz and high frequency stimulation of the STN
  Interventions: Device: 1 : S-C1-C2; Device: 2 : S-C2-C1; Device: 3 : C1 - S - C2; Device: 4 : C1 -C2 - S; Device: 5 : C2 - S - C1; Device: 6 : C2 - C1 - S

INTERVENTIONS:
Device: 1 : S-C1-C2 — Deep brain stimulation of the substantia nigra pars reticulata and of the subthalamic nucleus according to the order of randomisation (see intervention name) :
  * Standard stimulation
  * 125Hz at both STN and SNr for C1,
  * 125Hz for STN and 60 for SNr for C2
Device: 2 : S-C2-C1 — Deep brain stimulation of the substantia nigra pars reticulata and of the subthalamic nucleus according to the order of randomisation (see intervention name) :
  * Standard stimulation
  * 125Hz at both STN and SNr for C1,
  * 125Hz for STN and 60 for SNr for C2
Device: 3 : C1 - S - C2 — Deep brain stimulation of the substantia nigra pars reticulata and of the subthalamic nucleus according to the order of randomisation (see intervention name) :
  * Standard stimulation
  * 125Hz at both STN and SNr for C1,
  * 125Hz for STN and 60 for SNr for C2
Device: 4 : C1 -C2 - S — Deep brain stimulation of the substantia nigra pars reticulata and of the subthalamic nucleus according to the order of randomisation (see intervention name) :
  * Standard stimulation
  * 125Hz at both STN and SNr for C1,
  * 125Hz for STN and 60 for SNr for C2
Device: 5 : C2 - S - C1 — Deep brain stimulation of the substantia nigra pars reticulata and of the subthalamic nucleus according to the order of randomisation (see intervention name) :
  * Standard stimulation
  * 125Hz at both STN and SNr for C1,
  * 125Hz for STN and 60 for SNr for C2
Device: 6 : C2 - C1 - S — Deep brain stimulation of the substantia nigra pars reticulata and of the subthalamic nucleus according to the order of randomisation (see intervention name) :
  * Standard stimulation
  * 125Hz at both STN and SNr for C1,
  * 125Hz for STN and 60 for SNr for C2

SUMMARY:
The study is a pilot study on Parkinson's disease patients to evaluate Combined deep brain stimulation of the substantia nigra pars reticulata and of the subthalamic nucleus for unresponsive freezing of gait.

DETAILED DESCRIPTION:
One of the most challenging and unresolved problems in Parkinson's disease (PD) is the treatment of gait disorders, unresponsive to dopaminergic medication. Additionally, PD patients suffering from severe/unresponsive gait disorders are not considered good candidates for subthalamic nucleus deep brain stimulation (STN-DBS). Currently, there are no specific therapies to treat gait disorders in PD with an insufficient response to dopaminergic treatment. Furthermore, axial symptoms develop during disease progression even in operated patients. Axial symptoms are often one of the main causes of disability. There is evidence suggesting that low-frequency (LF) stimulation of the ventral area of the STN can improve axial symptoms. At the same time, the substantia nigra pars reticulata (SNr) is one of the most important output centers of the basal ganglia and is integrated within the locomotor control systems. Neurons within the SNr may act as high-frequency (HF) pacemakers, disrupting normal behavior downstream in the circuit. HF-STN in combination with LF or HF-SNr stimulation have been shown some beneficial effect on freezing of gait (FoG) among PD patients who had FoG unresponsive to dopaminergic therapy. However, only small pilot trials and case series have been investigated this strategy and evidences are scarce.

The aim of this study is to evaluate the effect of combined (C) stimulation of the STN and SNr on FoG if compared to standard (S) stimulation of the STN at 130 Hz, over one month. Based on previous literature evidence as primary aim the respective effect of two setting of C-stimulation will be separately assessed: a) C1- stimulation, with HF stimulation of the STN and SNr using a 'interleaved pulses' at 125 Hz vs. S- stimulation, over one month; b) C2-stimulation with LF stimulation of the SNr at 60Hz and HF stimulation of the STN vs. S- stimulation, over one month.

Other objectives are to evaluate the:

* Tolerance of combined stimulation (STN + SNr) through the collection of adverse events (AEs)
* Development of psychic events such as the presence of depression or dysphoria
* Effect of C (C1 and C2) -stimulation on walking disorders and other axial symptoms if compared vs. the S-stimulation.
* Effect of C (C1 and C2) -stimulation on PD's motor symptoms and motor complications if compared vs. the S-stimulation.
* Effect of C (C1 and C2) -stimulation on sleep quality if compared vs. the S-stimulation.

Each patient will have the 3 types of stimulation:

1. One month of S-stimulation (130hz, STN).
2. One month of C1- stimulation;
3. One month of C2- stimulation;

Stimulation setting order will be randomly assigned. Minimal dopaminergic treatment adjustment will be allowed to minimize the drop-out rate (± 100 mg of levodopa equivalent daily dose) and registered

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic PD defined as by the MDS Criteria ;
2. Patients submitted to STN-DBS, for at least 6 months;
3. Patients with STN-DBS at 130Hz;
4. Patients with a troublesome FoG according to the "NFOG-Q", Part II Item II ≥ 2 or Part III Item 7 ≥ 2;
5. Mini Mental State (MMS) ≥ 25 ;
6. Ventral contact of electrodes implanted in the SNr (according to analysis of activated tissue volume models (VTA));
7. Patients with stable parkinsonian stimulation parameters and anti-parkinsonian treatments for one month before the inclusion visit;
8. Patients with H/Y stage ≤ 3 in the Med ON/Stim On condition (at 130Hz, S-stimulation);

Exclusion Criteria:

1. Patient with atypical Parkinsonian syndrome;
2. Patient with severe FoG before DBS, i.e. MDS-UPDRS item 2.13 in Med ON ≥2 or MDS-UPDRS item 3.11 ≥2 in Med On;
3. Patient whose antiparkinsonian treatments were modified during the last month before inclusion;
4. Patient with H&Y stage ≥4 in Med On/Stim On (at 130Hz, S-stimulation) ;

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Score change of the " New freezing of gait questionnaire " | ONE MONTH AFTER INCLUSION
  the score change of the means of the New freezing of gait questionnaire at the end of each combined C1 and C2 stimulation, compared to S stimulation at one month of each period. The NFOG-Q is a clinician rated instrument used to evaluate FOG severity in patients with PD, unrelated to falls. Item responses use a 5-point scale ranging from 0 (absence of symptom) to 4 (severe). Total score ranges from 0 to 28; higher scores correspond to more severe FOG. Answers are based on experience over the past week or overall FOG during an entire day.

CONTACTS AND LOCATIONS:
Overall Officials: Margherita FABBRI, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Uh Toulouse, Toulouse, France

REFERENCES:
- [Background] Artusi CA, Ledda C, Gallo S, Rinaldi D, Campisi C, Rousseau V, Thalamas C, Barbosa R, Ory-Magne F, Brefel-Courbon C, Rascol O, de Barros A, Harroch E, Zibetti M, Rizzone MG, Romagnolo A, Imbalzano G, Lopiano L, Houeto JL, Fabbri M. Subthalamic and nigral stimulation for freezing of gait in Parkinson's disease: Randomized pilot trial. J Parkinsons Dis. 2024 Nov;14(8):1602-1613. doi: 10.1177/1877718X241292315. Epub 2025 Jan 17. PMID 39957196